CLINICAL TRIAL: NCT01037400
Title: Further Development of a Biochemical Approach to Measuring Surgical Trauma to Musculoskeletal Tissues
Brief Title: Biochemical Approach to Measuring Surgical Trauma
Status: Withdrawn | Type: Observational
Why Stopped: No patients recruited
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Anthony Adili, Associate Professor, McMaster University
Organization: McMaster University (Other)
Other Study IDs: TKR Study
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Total Knee Replacement
Keywords: Knee Replacement; Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total Knee Replacement Patients: Forty men and women ages 18-75 undergoing unilateral (n = 20) or bilateral (n = 20) knee replacement surgery with no musculoskeletal injury requiring medical attention in the past 3 months or producing pain in the previous 2 weeks and no inflammatory disease other than osteoarthritis.

SUMMARY:
This study will examine the magnitude and time course of changes in circulating (serum and plasma) biomarker concentrations associated with musculoskeletal injury created by total knee replacement surgery. The sensitivity to injury will be characterized by the changes in mean serum concentration before and after surgery. Specificity for the injured state will be evaluated comparing the baseline to peak change (injury response) with the pre-surgery to follow-up baseline fluctuation (i.e. measurement noise).

ELIGIBILITY:
Inclusion Criteria

* Age 18 to 75
* No musculoskeletal injury requiring medical attention in the past 3 months other than entirely related to worsening symptoms of the operative knee or spinal level.
* No musculoskeletal injury producing pain in the previous 2 weeks.
* No inflammatory disease other than osteoarthritis)
* No exercise with weights in the 2 weeks before surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Forty men and women ages 18-75 undergoing unilateral (n = 20) or bilateral (n = 20) knee replacement surgery with no musculoskeletal injury requiring medical attention in the past 3 months or producing pain in the previous 2 weeks and no inflammatory disease other than osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of biomarkers in response to tissue injury | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare, Hamilton, Ontario, Canada